CLINICAL TRIAL: NCT03927573
Title: A Multicenter, Open-label, Dose-escalating, Phase I Trial With GEM3PSCA, a PSCA Targeted Bispecific Antibody Engaging T-cells, in Patients With Progressive Disease After Standard Systemic Therapy in Cancers With Positive PSCA Marker
Brief Title: Study With Bispecific Antibody Engaging T-cells, in Patients With Progressive Cancer Diseases With Positive PSCA Marker
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: business decision by sponsor
Sponsor: AvenCell Europe GmbH (Industry)
Collaborators: GCP-Service International Ltd. & Co. KG (Industry)
Responsible Party: Sponsor
Organization: AvenCell Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GEM3PSCA-01
Record Dates: First submitted 2019-04-16; First posted 2019-04-25 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Non-small Cell Lung Cancer; Prostate Cancer; Renal Cancer; Transitional Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms; Kidney Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: Dose escalation scheme; Single patient cohorts on the first three dose levels, 3+3 afterwards.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GEM3PSCA (Experimental): Application of GEM3PSCA, a PSCA targeted bispecific antibody engaging T-cells
  Interventions: Drug: GEM3PSCA

INTERVENTIONS:
Drug: GEM3PSCA — Infusion of GEM3PSCA, administered intravenously, continuously over 7 days, 2 cycles

SUMMARY:
This dose-escalating phase I trial assesses for the first time the safety, the side effects and the harmlessness, as well as the therapeutical benefit of the new study drug GEM3PSCA in patients with prostate stem cell antigen (PSCA) expressing cancer types which failed to respond to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, ≥ 18 years of age
2. Progressive PSCA positive cancer (urogenital tract (renal, transitional cell, prostate), non-small cell lung) refractory to standard treatments and with no other available standard or curative treatment
3. Measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
5. Life expectancy of at least 2 months
6. Platelets > 50,000/µl
7. Hemoglobin > 9 g/dl
8. Adequate renal and hepatic laboratory assessments
9. Adequate pulmonary function with oxygen saturation (SpO2) ≥ 90 % and no structural pulmonary disease which might jeopardize patient safety according to judgement of the investigator
10. Left ventricular ejection fraction (LVEF) of ≥ 45 %
11. Existing port-system or central venous catheter resp. acceptance of implantation of a device
12. A female of childbearing potential may be enrolled providing she has a negative pregnancy test at screening visit and is routinely using a highly effective method of birth control resulting in a low failure rate (e.g. hormonal contraception, intrauterine device, total sexual abstinence or sterilization) until 3 months from the last study drug administration. Male patients must also practice a highly effective method of birth Control
13. Able to give written informed consent

Exclusion Criteria:

1. Other malignancy requiring active therapy
2. Non-measurable tumor disease
3. Patients with active brain metastases (patients with brain metastases or residue after resection with stable size for 6 months in MRI not older than 8 weeks, after consultation with the sponsor, are not excluded from the trial)
4. Use of chemotherapy and radiotherapy within 2 weeks prior to start of trial medication
5. Use of checkpoint inhibitors (having a marketing authorization) within a washout of 5 x t1/2 (half-life); patients with experimental checkpoint inhibitors at all
6. Other investigational drug within the past 4 weeks before start of trial medication
7. Patients undergoing renal dialysis
8. Pulmonary disease with clinical relevant hypoxia
9. Evidence of active, non-infectious pneumonitis or history of interstitial lung disease
10. Cardiac disease: i.e. heart failure NYHA (New York Heart Association) III or IV, unstable coronary artery disease
11. Active central nervous disease (e.g. Parkinson, multiple sclerosis, seizures) and stroke within last 6 months
12. Active gastrointestinal ulceration or bleeding within the last 6 months unless related to underlying malignant disease
13. Renal outflow obstruction, macroscopic or significant microscopic hematuria
14. Active infectious diseases considered by investigator to be incompatible with protocol
15. Major surgery within 28 days
16. Autoimmune diseases requiring steroids at a dose above 10 mg prednisolone equivalent or other immunosuppressants
17. Pregnant or breastfeeding women
18. Psychiatric disorders, drug and/or alcohol abuse
19. Known history of human immunodeficiency virus (HIV) or active/chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV)
20. Known hypersensitivity to GEM3PSCA excipients
21. Evidence suggesting that the patient is not likely to follow the study protocol (e.g. lacking compliance)
22. Incapability of understanding purpose and possible consequences of the trial
23. Patients who should not be included according to the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | End of Treatment (EOT) +14 days (DLT period)
  MTD is the previous dose level of the cohort where a DLT is observed in at least wo subjects.
Incidence and intensity of adverse events | End of Treatment (EOT) +14 days (DLT period)
  graded according to CTCAE V4.03
Incidence of Dose limiting toxicity (DLT) | End of Treatment (EOT) +14 days (DLT period)
  Dose Limiting Toxicity is defined as any event at least possibly related to investigational medicinal product (IMP)

SECONDARY OUTCOMES:
Recommended phase 2 dose (RP2D) | From start of treatment until up to 14 days after last treatment cycle (2 initial cycles + max. 6 additional cycles per patient). Each cycle consists of 7 days treatment plus DLT evaluation period (14 days)
  The RP2D will be determined based on MTD, all available efficacy data, and all available safety data, including information derived from additional treatment cycles.
Antitumor activity of GEM3PSCA according to RECIST1.1 (Response Evaluation Criteria in Solid Tumors) | End of Treatment (EOT) +14 days (DLT period)
  response rates
Prostate specific antigen (PSA) response in patients with prostate cancer | End of Treatment (EOT) +14 days (DLT period)
Overall survival (OS) | End of Treatment (EOT) + 14 days (DLT period)
Influence on circulating tumor cells in patients with prostate cancer | Day 8 / End of Treatment (EOT)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Bargou, Prof. Dr., Principal Investigator — Universitätsklinikum Würzburg, Interdisziplinäres Studienzentrum mit ECTU
Locations (5):
- Germany (5):
  - Klinikum rechts der Isar der TU München, Munich, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Marburg, Marburg, Hesse
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No